CLINICAL TRIAL: NCT02374827
Title: Complete Salpingectomy Versus Standard Postpartum Tubal Ligation at the Time of Cesarean Delivery- a Randomized Controlled Study
Brief Title: Salpingectomy at Cesarean Delivery for Ovarian Cancer Reduction (SCORE)
Acronym: SCORE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Akila Subramaniam, MD, Maternal-Fetal Medicine Fellow, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: F140630003 (ST)
Record Dates: First submitted 2015-02-23; First posted 2015-03-02 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-10

CONDITIONS: Ovarian Cancer
Keywords: complete salpingectomy; standard tubal ligation; cesarean delivery; feasibility; safety; partial salpingectomy
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard postpartum tubal ligation (Active Comparator): In this arm, patients will receive the standard postpartum tubal ligation by accepted methods (procedure names are the following: Modified pomeroy technique or Parkland method). These methods are procedures for completing a partial salpingectomy.
  Interventions: Procedure: Standard postpartum tubal ligation
- Complete Salpingectomy (Experimental): In this arm, patients will receive a complete salpingectomy by documented accepted methods.
  Interventions: Procedure: Complete Salpingectomy

INTERVENTIONS:
Procedure: Standard postpartum tubal ligation — Patients will undergo a standard postpartum tubal ligation by accepted documented surgical procedural methods (Modified Pomeroy or Parkland method)
  Arms: Standard postpartum tubal ligation
Procedure: Complete Salpingectomy — Patients will undergo a complete salpingectomy by a documented surgical protocol established by accepted surgical procedural methods.
  Arms: Complete Salpingectomy

SUMMARY:
To compare the feasibility and surgical outcomes between complete salpingectomy and standard postpartum tubal ligation (partial salpingectomy) at the time of cesarean delivery in women with undesired future fertility. as a possible ovarian cancer risk-reducing procedure.

DETAILED DESCRIPTION:
All pregnant women receiving prenatal care within the UAB Health System, and planning to undergo tubal ligation at the time of their scheduled cesarean delivery (primary or repeat) will be approached about the study. Patients will be randomized to receive either the standard tubal ligation practice at our institution (modified Pomeroy procedure or Parkland) or a complete salpingectomy. The objective of this trial is to evaluate if a complete salpingectomy can be performed safely and comparable to a standard postpartum tubal ligation.

ELIGIBILITY:
Inclusion Criteria:

* All pregnant women > 25 years receiving prenatal care within the UAB Health System, and planning to undergo tubal ligation at the time of their scheduled cesarean delivery (primary or repeat)
* Informed consent obtained

Exclusion Criteria:

* Inability to obtain informed consent
* Fetal death or anomalies
* Preterm delivery < 36 weeks gestation
* Immune-compromising disease
* Chronic steroid use
* Chronic prophylactic or therapeutic anti-coagulation
* Patients no followed in our regional health system
* Known BRCA mutation carrier status
* Age < 25 years

Min Age: 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Time to complete sterilization procedure | At time of procedure
  The primary outcome will involve measuring the amount of surgical time required to complete the assigned sterilization procedure
Completion rate of sterilization procedure | At time of procedure
  The primary outcome will involve assessing the completion rate of assigned sterilization procedure

SECONDARY OUTCOMES:
Total operative time | At time of procedure
  Includes cesarean delivery and sterilization procedure time
Mean post-operative pain score | Postpartum admission (3-4 days)
Perioperative complication rate | From time of procedure to 6 weeks postpartum
  Composite assessment of the following: estimated blood loss, need for blood transfusion, intra-abdominal hemorrhage/hematoma, need for readmission, need for reoperation, need for additional surgical procedure, major post-operative complication

CONTACTS AND LOCATIONS:
Overall Officials: Akila Subramaniam, MD, MPH, Principal Investigator — University of Alabama at Birmingham; Britt K Erickson, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Ostby SA, Blanchard CT, Sanjanwala AR, Szychowski JM, Leath CA 3rd, Huh WK, Subramaniam A. Feasibility, Safety, and Provider Perspectives of Bipolar Electrosurgical Cautery Device for (Opportunistic or Complete) Salpingectomy at the Time of Cesarean Delivery. Am J Perinatol. 2024 Apr;41(6):804-813. doi: 10.1055/s-0042-1748525. Epub 2022 Jun 21. PMID 35728603
- [Derived] Subramaniam A, Einerson BD, Blanchard CT, Erickson BK, Szychowski J, Leath CA 3rd, Biggio JR, Huh WK. The cost-effectiveness of opportunistic salpingectomy versus standard tubal ligation at the time of cesarean delivery for ovarian cancer risk reduction. Gynecol Oncol. 2019 Jan;152(1):127-132. doi: 10.1016/j.ygyno.2018.11.009. Epub 2018 Nov 23. PMID 30477808
- [Derived] Subramaniam A, Blanchard CT, Erickson BK, Szychowski J, Leath CA, Biggio JR, Huh WK. Feasibility of Complete Salpingectomy Compared With Standard Postpartum Tubal Ligation at Cesarean Delivery: A Randomized Controlled Trial. Obstet Gynecol. 2018 Jul;132(1):20-27. doi: 10.1097/AOG.0000000000002646. PMID 29889762